CLINICAL TRIAL: NCT01871493
Title: A Phase 1 Study to Evaluate the Pharmacokinetics of LY2605541 Injection and Insulin Lispro Injection Administered as Mixture or as Individual Components in Healthy Subjects
Brief Title: A Study of LY2605541 and Insulin Lispro Mixture in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14833; I6O-FW-BHBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY2605541; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- LY2605541-Part A (Experimental): 1.42 units per kilogram (U/kg) of LY2605541 given once daily (QD) for 1 day, subcutaneously (SQ) in 1 of 4 treatment periods.
  Interventions: Drug: LY2605541
- Insulin Lispro-Part A (Active Comparator): Single dose 0.36 U/kg of insulin lispro given QD for 1 day, SQ in 1 of 4 treatment periods.
  Interventions: Drug: Insulin Lispro
- LY2605541/Lispro Mix 1-Part A (Experimental): Single dose 0.54 U/kg of LY2605541 and 0.36 U/kg insulin lispro mixture given QD for 1 day, SQ in 1 of 4 treatment periods.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro
- LY2605541/Lispro Mix 2-Part A (Experimental): Single dose 1.42 U/kg of LY2605541 and 0.36 insulin lispro mixture given QD for 1 day, SQ in 1 of 4 treatment periods.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro
- Insulin Lispro-Part B (Active Comparator): 0.18 U/kg insulin lispro given twice daily (BID) for 1 day, SQ in 1 of 4 treatment periods. Part B is contingent on data from Part A.
  Interventions: Drug: Insulin Lispro
- LY2605541/Lispro Mix-Part B (Experimental): 0.71 U/kg LY2605541 and 0.18 U/kg insulin lispro mixture given BID for 1 day, SQ in 1 of 4 treatment periods. Part B is contingent on data from Part A.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro
- LY2605541 QD-Part B (Experimental): 0.54 U/kg of LY2605541 given QD for 1 day, SQ in 1 of 4 treatment periods. Part B is contingent on data from Part A.
  Interventions: Drug: LY2605541
- LY2605541 BID-Part B (Experimental): 0.71 U/kg of LY2605541 given BID for 1 day SQ in 1 of 4 treatment periods. Part B is contingent on data from Part A.
  Interventions: Drug: LY2605541

INTERVENTIONS:
Drug: LY2605541 — Administered subcutaneous (SQ)
  Arms: LY2605541 BID-Part B; LY2605541 QD-Part B; LY2605541-Part A; LY2605541/Lispro Mix 1-Part A; LY2605541/Lispro Mix 2-Part A; LY2605541/Lispro Mix-Part B
Drug: Insulin Lispro — Administered SQ
  Other Names: Humalog
  Arms: Insulin Lispro-Part A; Insulin Lispro-Part B; LY2605541/Lispro Mix 1-Part A; LY2605541/Lispro Mix 2-Part A; LY2605541/Lispro Mix-Part B

SUMMARY:
The main purpose of this study is to evaluate how the body absorbs and removes LY2605541, insulin lispro, and a mixture of both from the blood. The study has two parts. Participants may enroll in only one part. Each part has four treatment periods in a fixed order. The study will last approximately 8 weeks, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are not of child-bearing potential
* Have a body mass index (BMI) between 18 and 29.9 kilograms per meter squared (kg/m^2), inclusive
* Are nonsmokers or have not smoked for at least 2 months prior to entering the study

Exclusion Criteria:

* Have known allergies to insulin or its excipients, or related drugs, or history of relevant allergic reactions of any origin
* Have a history of first-degree relatives known to have diabetes mellitus
* Have used systemic glucocorticoids within 3 months prior to entry into the study
* Have donated blood or had a blood loss of 450 milliliter (mL) within 1 month prior to study enrollment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Time to Reach Peak Concentration (tmax) of LY2605541 and Insulin Lispro | Pre-dose up to 216 hours post-dose
Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY2605541 and Insulin Lispro | Pre-dose up to 216 hours post-dose
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-∞) of LY2605541 and Insulin Lispro | Pre-dose up to 216 hours post-dose

SECONDARY OUTCOMES:
Maximum Glucose Infusion Rate (Rmax) | Predose up to 32 hours post clamp procedure in all treatment periods
Total Glucose Infused Over Clamp Duration (Gtot) | Predose up to 32 hours post clamp procedure in all treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore